CLINICAL TRIAL: NCT00986830
Title: Healthcare Utilization and Outcomes of FinESS Treatment in the Office
Acronym: RELIEF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Entellus Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1630-001
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Results first posted 2020-10-27 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Rhinosinusitis
Keywords: Rhinosinusitis; Balloon catheters; Office treatment; Otorhinolaryngologic diseases; Respiratory tract infections; Respiratory tract diseases; FinESS Sinus Treatment; Endoscopic sinus surgery
MeSH Terms: conditions — Rhinosinusitis; Otorhinolaryngologic Diseases; Respiratory Tract Infections; Respiratory Tract Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

ARMS (1):
- Balloon Dilation (Experimental): Balloon dilation of the maxillary sinuses using the FinESS Sinus Treatment device.
  Interventions: Device: FinESS Sinus Treatment

INTERVENTIONS:
Device: FinESS Sinus Treatment

SUMMARY:
A prospective, nonrandomized trial to evaluate postoperative healthcare resource utilization after maxillary balloon antrostomy using FinESS Sinus Treatment in the physician's office.

DETAILED DESCRIPTION:
A prospective, nonrandomized trial to evaluate postoperative healthcare resource utilization after maxillary balloon antrostomy using FinESS Sinus Treatment in the physician's office. Also to demonstrate the long-term durability of FinESS Sinus Treatment performed in an office setting.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Male or female subjects
* Diagnosis of rhinosinusitis (CT radiographic evidence and medical evaluation)
* Willing to comply with protocol requirements
* Able to provide consent

Exclusion Criteria:

* Hemophilia
* Cystic fibrosis
* Ciliary dysfunction
* Severe septal deviation causing obstruction of the ostiomeatal unit
* Pregnant females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2009-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Central California ENT, Fresno, California
  - South Denver ENT and Allergy, Denver, Colorado
  - ENT and Allergy Associates, Trumbull, Connecticut
  - NorthShore University, Evanston, Illinois
  - Advanced ENT and Allergy, Louisville, Kentucky
  - St. Cloud Ear, Nose and Throat, Saint Cloud, Minnesota
  - Coastal Ear, Nose and Throat Associates, New Bern, North Carolina
  - Midwest Ear, Nose and Throat, Sioux Falls, South Dakota
  - Holston Medical Center, Kingsport, Tennessee
  - Austin Ear, Nose and Throat, Austin, Texas
  - Texas Sinus Center, Boerne, Texas
  - The Snoring Center, Dallas, Texas
  - Advanced Otolaryngology PC, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Levine SB, Truitt T, Schwartz M, Atkins J. In-office stand-alone balloon dilation of maxillary sinus ostia and ethmoid infundibula in adults with chronic or recurrent acute rhinosinusitis: a prospective, multi-institutional study with-1-year follow-up. Ann Otol Rhinol Laryngol. 2013 Nov;122(11):665-71. doi: 10.1177/000348941312201101. PMID 24358625

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Balloon Dilation
Started | 74
Treated | 69
Completed | 66
Not Completed | 8
Not completed — Death | 1
Not completed — Lost to Follow-up | 1
Not completed — Lack of Efficacy | 1
Not completed — Unable to access sinus with device | 5

BASELINE CHARACTERISTICS:
Population: All enrolled participants treated with the FinESS Sinus Treatment device.
Arm/Group | Balloon Dilation
Number analyzed (Participants) | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.1 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 25
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 69
Previous sinus surgery [Count of Participants; unit: Participants] | 7
Affected sinuses [Count of Participants; unit: Participants]
  Maxillary only | 55
  Maxillary and anterior ethmoid | 14

OUTCOME MEASURES:

1. Primary Outcome: Sino-Nasal Outcomes Test
Description: The 20-item Sino-Nasal Outcomes Test (SNOT-20) is a validated, disease-specific patient-reported instrument designed to indicate the severity of rhinosinusitis symptoms. The SNOT-20 evaluates 20 symptoms on a scale from 0 ("no problem") to 5 ("problem as bad as it can be"). The overall SNOT-20 score is the average of the 20 symptoms scores providing a range from 0 to 5 with higher scores indicating worse symptoms. The minimal clinically important difference (MCID) has been determined to be a reduction of 0.8 or more in the overall SNOT-20 score.
Time Frame: Baseline and 12 months post procedure
Population: All treated participants with baseline and 12-month SNOT-20 scores.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Balloon Dilation
Number analyzed (Participants) | 64
score on a scale
  Baseline | 2.3 (0.9)
  12-Month follow-up | 1.1 (1.0)
Statistical Analysis 1: Comparison: Balloon Dilation; Test type: Superiority; p < 0.0001, t-test, 2 sided — Paired t-tests were used to calculate the p-values and evaluate whether the change in outcomes from baseline to follow-up were statistically different from zero. A p value of <0.05 was considered statistically significant; A reduction in SNOT-20 score of 0.8 or more is considered clinically meaningful

2. Secondary Outcome: Rhinosinusitis Symptom Inventory (RSI) Nasal Symptoms Domain
Description: The Rhinosinusitis Symptom Inventory (RSI) is a self-administered quality of life questionnaire. Section 1 of the questionnaire scores symptoms related to chronic rhinosinusitis on a 6-point scale with "0" indicating no symptoms and "5" indicating very severe symptoms. There are 4 symptoms domains: nasal, facial, oropharyngeal, and systemic. RSI domain scores are calculated by summing the score of the specific domain question, dividing by the number of domain questions, and multiplying by 20 to obtain a standardized score. Scores can range from 0 to 100 with higher scores indicating worse symptoms.
Time Frame: Baseline and 12 months post procedure
Population: All treated participants with baseline and 12-month RSI scores.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Balloon Dilation
Number analyzed (Participants) | 65
score on a scale
  Baseline | 53.7 (23.9)
  12-Month Follow-up | 20.7 (21.1)
Statistical Analysis 1: Comparison: Balloon Dilation; Test type: Superiority; p < 0.0001, t-test, 2 sided — Paired t-tests were used to calculate the p-values and evaluate whether the change in outcomes from baseline to follow-up were statistically different from zero. A p value <0.05 is considered statistically significant

3. Secondary Outcome: Rhinosinusitis Symptom Inventory (RSI) Facial Symptoms Domain
Description: as for outcome 2
Time Frame: Baseline and 12 months post procedure
Population: All treated participants with baseline and 12-month RSI scores.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Balloon Dilation
Number analyzed (Participants) | 65
score on a scale
  Baseline | 61.4 (24.0)
  12-Month Follow-up | 24.4 (23.9)
Statistical Analysis 1: Comparison: Balloon Dilation; Test type: Superiority; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 2, analysis 1]

4. Secondary Outcome: Rhinosinusitis Symptom Inventory (RSI) Oropharyngeal Symptoms Domain
Description: as for outcome 2
Time Frame: Baseline and 12 months post procedure
Population: All treated participants with baseline and 12-month RSI scores.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Balloon Dilation
Number analyzed (Participants) | 65
score on a scale
  Baseline | 40.6 (20.3)
  12-Month Follow-up | 15.4 (15.9)
Statistical Analysis 1: Comparison: Balloon Dilation; Test type: Superiority; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 2, analysis 1]

5. Secondary Outcome: Rhinosinusitis Symptom Inventory (RSI) Systemic Symptoms Domain
Description: as for outcome 2
Time Frame: Baseline and 12 months post procedure
Population: All treated participants with baseline and 12-month RSI scores.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Balloon Dilation
Number analyzed (Participants) | 65
score on a scale
  Baseline | 40.6 (22.4)
  12-Month Follow-up | 15.4 (18.6)
Statistical Analysis 1: Comparison: Balloon Dilation; Test type: Superiority; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 2, analysis 1]

6. Secondary Outcome: Number of Participants Using Nasal Steroids
Description: The Rhinosinusitis Symptom Inventory (RSI) is a self-administered quality of life questionnaire. Section 2 of the questionnaire records medication usage (nasal steroid sprays, anti-histamines, and antibiotics) over the past 12 months.
Time Frame: Baseline and 12 months post procedure
Population: All treated participants with baseline and 12-month RSI scores.
Measure: Count of Participants; unit: Participants
Arm/Group | Balloon Dilation
Number analyzed (Participants) | 65
Participants
  Baseline | 47
  12-Month Follow-up | 36
Statistical Analysis 1: Comparison: Balloon Dilation; Test type: Superiority; p = 0.009, t-test, 2 sided — Paired t-tests were used to calculate the p-values and evaluate whether the change in outcomes from baseline to follow-up were statistically different from zero. A p value <0.05 indicates statistical significance

7. Secondary Outcome: Number of Participants Using Antihistamines
Description: as for outcome 6
Time Frame: Baseline and 12 months post procedure
Population: All treated participants with baseline and 12-month RSI scores.
Measure: Count of Participants; unit: Participants
Arm/Group | Balloon Dilation
Number analyzed (Participants) | 65
Participants
  Baseline | 33
  12-Month Follow-up | 28
Statistical Analysis 1: Comparison: Balloon Dilation; Test type: Superiority; p = 0.292, t-test, 2 sided — [p-value comment as in outcome 6, analysis 1]

8. Secondary Outcome: Number of Participants Using Antibiotics
Description: as for outcome 6
Time Frame: Baseline and 12 months post procedure
Population: All treated participants with baseline and 12-month RSI scores. Four participants with blank responses at either interval are considered not evaluable.
Measure: Mean (Standard Deviation); unit: number of antibiotic courses
Arm/Group | Balloon Dilation
Number analyzed (Participants) | 61
number of antibiotic courses
  Baseline | 5.5 (2.5)
  12-Month Follow-up | 2.3 (2.4)
Statistical Analysis 1: Comparison: Balloon Dilation; Test type: Superiority; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 6, analysis 1]

9. Secondary Outcome: Number of Participants With Device and/or Procedure-related Adverse Events
Description: Number of participants with 1 or more adverse events considered possibly or definitely related to the FinESS device and/or balloon dilation procedure.
Time Frame: Baseline through 12 months post procedure
Population: All enrolled participants. Participants with unsuccessful procedures (sinus could not be accessed and dilated) were followed for 1 week post procedure. Treated participant are evaluated through 12 months post procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | Balloon Dilation
Number analyzed (Participants) | 74
Participants | 16

ADVERSE EVENTS:
Time Frame: 12 months post procedure for treated participants. Participants with unsuccessful treatment were followed for 1 week post procedure.
Description: Adverse event information was collected on a standardized case report form at each follow-up visit.
Arm/Group | Balloon Dilation
All-Cause Mortality (participants affected / at risk) | 1/74
Serious Adverse Events (participants affected / at risk) | 0/74
Other Adverse Events (participants affected / at risk) | 9/74
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Balloon Dilation (N=74)
Numbness (Injury, poisoning and procedural complications) | 9 (9) — Mild numbness in the treatment area (face, cheek, lip, teeth, eye)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days